CLINICAL TRIAL: NCT05606237
Title: Efficacy of Repeated Low-level Red-light Therapy in Myopia Control: a Single Arm Controlled Trial
Brief Title: Efficacy of Repeated Low-level Red-light Therapy in Myopia Control
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: University of Melbourne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-35793
Record Dates: First submitted 2022-09-21; First posted 2022-11-04 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Myopia
Keywords: myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Intervention Model Description: This trial is a single-center, multi-ethnic, single-blind, single arm controlled trial designed to evaluate the efficacy and safety of low level red light treatment on myopia among multi-ethnic schoolchildren.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Low Level Red Light Treatment Arm (Experimental): On top of wearing single vision spectacles, subjects in the intervention group will receive low-level red light treatment twice a day from Monday to Friday, with each treatment lasting for 3 minutes at a minimal interval of 4 hours.
  Interventions: Device: Low-level Red Light Therapy Device

INTERVENTIONS:
Device: Low-level Red Light Therapy Device — The treatment device used in this study is a semi-conductor laser product (Eyerising International Pty Ltd, Melbourne, Australia), emitting low-level red-light with a wavelength of 650 ± 10 nm. Based on calculations done by the manufacturer, the device provides light at a power of 2.00 ± 0.50 mW.

SUMMARY:
Low-level red-light technology provides a new and innovative myopia control approach. This strategy enables relatively high energies of light to be delivered at much shorter durations of exposure to induce the myopia control effect. The efficacy of the low-level red-light technology has been proven in a Chinese population. This trial demonstrated that 3-minutes per session twice a day repeated low-level red-light treatment controlled 87.7% of refraction progression and 76.8% of axial length elongation when the time of compliance to the treatment was 75%. Repeating this RCT in culturally diverse groups will confirm and translate this technology into a solution for myopia control globally.

DETAILED DESCRIPTION:
The purpose of this study is to assess the safety and efficacy of low level red light therapy in myopia control in African, Hispanic, and Caucasian children. This is a prospective, multi-ethnic, parallel-controlled randomized trial that will enroll myopic children aged 8-13 years old as subjects. On top of wearing single vision spectacles, subjects in the intervention group will receive treatment twice a day from Monday to Friday, with each treatment lasting for 3 minutes at a minimal interval of 4 hours. Subjects in the control group will wear single vision spectacles. The study will evaluate axial elongation, cycloplegic spherical equivalent change, changes in other biological parameters (except axial length), and uncorrected and best corrected visual acuity of the two groups of subjects at 1 month, 3 months, 6 months, and 12 months after enrollment. The study plans to conduct an interim analysis at a three-month follow-up. The enrollment target is 90 participants: 30 Hispanic Children (15 control and 15 treatment) , 30 African Children (15 control and 15 treatment), and 30 Caucasian Children (15 control and 15 treatment).

ELIGIBILITY:
Inclusion Criteria:

1. Provision of consent
2. Non-Chinese Ethnicity
3. Age: ≥8 and ≤13 years at enrollment
4. Myopia: Spherical equivalent refractions (SERs) under cycloplegia: -1.00 to -5.00 diopters (D)

4) Astigmatism of 2.50 D or less 5) Anisometropia of 1.50 D or less 6) Corrected monocular logMAR visual acuity (VA): 1.0 or better 7) Consent to participate in random allocation of grouping 8) Fluent in English 9) Willing and able to participate in all required activities of the study6) Corrected monocular logMAR visual acuity (VA): 1.0 or better

Exclusion Criteria:

1. Strabismus and binocular vision abnormalities in either eye
2. Ocular abnormalities in either eye or other systemic abnormalities that affect participate in all required activities of the study.
3. Other reasons, including but not limited to severe physical and cognitive disability, that the physician may consider inappropriate for enrollment
4. Noncompliance with treatment
5. Children whose parents do not sign informed consent

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2023-07-14 (Actual); Primary Completion 2027-01-14 (Estimated); Study Completion 2027-01-14 (Estimated)

PRIMARY OUTCOMES:
Axial Length (AL) (mm) at Baseline | 1 month
  Axial Length (AL) is characterized as the combination of anterior chamber depth, lens thickness and vitreous chamber depth and measured by results from the IOLMaster. AL will be taken at the 1-, 3-, 6-, and 12-month follow-up visits.
Axial Length (AL) (mm) at Month 1 | 1 month
  Axial Length (AL) is characterized as the combination of anterior chamber depth, lens thickness and vitreous chamber depth and measured by results from the IOLMaster. AL will be taken at the 1-, 3-, 6-, and 12-month follow-up visits.
Axial Length (AL) (mm) at Month 3 | 3 months
  Axial Length (AL) is characterized as the combination of anterior chamber depth, lens thickness and vitreous chamber depth and measured by results from the IOLMaster. AL will be taken at the 1-, 3-, 6-, and 12-month follow-up visits.
Axial Length (AL) (mm) at Month 6 | 6 months
  Axial Length (AL) is characterized as the combination of anterior chamber depth, lens thickness and vitreous chamber depth and measured by results from the IOLMaster. AL will be taken at the 1-, 3-, 6-, and 12-month follow-up visits.
Axial Length (AL) (mm) at Year 1 | 1 Year
  Axial Length (AL) is characterized as the combination of anterior chamber depth, lens thickness and vitreous chamber depth and measured by results from the IOLMaster. AL will be taken at the 1-, 3-, 6-, and 12-month follow-up visits.

CONTACTS AND LOCATIONS:
Overall Officials: Tiffany Chen, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results after deidentification(text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Immediately following publication. No end date.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose. For individual participant data meta-analysis.

REFERENCES:
- [Background] Holden BA, Fricke TR, Wilson DA, Jong M, Naidoo KS, Sankaridurg P, Wong TY, Naduvilath TJ, Resnikoff S. Global Prevalence of Myopia and High Myopia and Temporal Trends from 2000 through 2050. Ophthalmology. 2016 May;123(5):1036-42. doi: 10.1016/j.ophtha.2016.01.006. Epub 2016 Feb 11. PMID 26875007

DOCUMENTS (2):
  • Study Protocol (2022-08-22): https://cdn.clinicaltrials.gov/large-docs/37/NCT05606237/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-22): https://cdn.clinicaltrials.gov/large-docs/37/NCT05606237/SAP_001.pdf